CLINICAL TRIAL: NCT06272526
Title: Acceptability and Effectiveness Study of Internet Based Social Anxiety Intervention for University Students in Turkey : A Randomized Controlled Trial
Brief Title: Internet-Based Self-Help Intervention for Social Anxiety Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anadolu University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOCIALANX_1
Record Dates: First submitted 2024-02-14; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Mental Health Issue
Keywords: Cognitive Behavioral Therapy; Web-based intervention; procrastation

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Web-Based Intervention (Experimental): Participants in this group will use the web-based intervention (https://kendikendineyardim.org) with guidance support.
  Interventions: Other: Internet Based Intervention - GUIDED
- Waitlist (No Intervention): The waiting list control group participants will be controlled for time and assessed during the first 7-week period. Participants will have no contact with the study team during the waiting period. Immediately after the waiting period, they will receive the internet-based intervention with the experimental group.

INTERVENTIONS:
Other: Internet Based Intervention - GUIDED — The experimental group participants will be in treatment through web-based intervention consisting of five to seven weeks. The intervention program will be offered to participants through the website https://kendikendineyardim.org, the online self-help platform in Turkey. Participants will be able to use the system with their e-mail addresses and passwords.The intervention consists of five modules consisting of behavioral, emotional and cognitive content. The modules include text, interactive forms, animated videos, audio recordings, and images. Participants in this arm will receive weekly feedback from guides via the platform's message sending feature.
  Arms: Guided Web-Based Intervention

SUMMARY:
This study is a randomized-controlled trial in which the assumed superiority of the module internet-based cognitive behavioral therapy intervention for social anxiety disorder is evaluated compared to a waitlist control group. Participants will be assigned to one of two groups, treatment which have web-based intervention (guided), and waitlist.

The intervention program will be offered to treatment group participants (guided) through the website https://kendikendineyardim.org, the unique online self-help platform in Turkey. Participants in the web-based treatment group will receive feedback message within 24 hours after each completed module from the guides.

DETAILED DESCRIPTION:
This study is a randomized-controlled trial in which the assumed superiority of the module internet-based cognitive behavioral therapy intervention for social anxiety disorder is evaluated compared to a waitlist control group. Participants will be assigned to one of two groups, treatment which have web-based intervention (guided), and waitlist.

The intervention program will be offered to treatment group participants (guided) through the website https://kendikendineyardim.org, the unique online self-help platform in Turkey. Participants in the web-based treatment group will receive feedback message within 24 hours after each completed module from the guides.

The intervention program consists of five modules. Each module can be completed in 30-40 minutes. Each module starts with the evaluation of the exercises given at the end of the previous module and ends with a between-module exercise. The module includes text, interactive forms, animated videos, audio recordings, and images.

The duration of the program will be approximately five to seven weeks. However, participants will be allowed to follow the program at their own speed. No limitations will be imposed other than the completion of no more than one module per day. Users can use the system with their e-mail addresses and passwords.

The data will be compared with suitable statistical techniques.

ELIGIBILITY:
Inclusion Criteria:

* volunteering to participate in the study;
* having a valid e-mail address;
* having internet access (computer, laptop, tablet, or mobile device);
* being aged 18 or older;
* score of 25 or above on both anxiety and avoidance subscales of the Liebowitz Social Anxiety Scale Turkish Form

Exclusion Criteria:

* receiving any psychological help (i.e., medication or psychotherapy/counseling) during the research period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale (LSAS) Turkish Form | Baseline, post-test (6 weeks later from baseline), follow up (10 weeks later from baseline)
  This scale, developed by Liebowitz (1987), aims to evaluate in which social situations individuals with social phobia encounter anxiety. It includes 24 items divided into two subscales addressing social interaction (11 items) and performance (13 items). Items are rated on a 4-point scale for anxiety. When looking at the scoring of the scale, the higher the individual scores, the more anxiety and avoidance behaviors they have. It is a self-report tool and participants evaluate themselves.

SECONDARY OUTCOMES:
Social Appearance Anxiety Scale (SAAS) Turkish Form | Baseline, post-test (6 weeks later from baseline), follow up (10 weeks later from baseline)
  It is a 5-point Likert type scale developed to measure an individual's emotional, behavioral and cognitive concerns about their appearance. The Turkish form of the scale consists of 16 items. The lowest total score from the scale is 16 and the highest score is 80. High scores indicate high social appearance anxiety. It is a self-report tool and participants evaluate themselves.
Patient Health Questionnaire-9 (PHQ-9) Turkish Form | Baseline, post-test (6 weeks later from baseline), follow up (10 weeks later from baseline)
  For asses depression symptoms level. PHQ-9 consists of 9 items structured on a four-point Likert scale (0-3) to measure the level of depressed mood. The lowest score is 0 and the highest score is 27. A high score indicates a high level of depression. It is a self-report tool and participants evaluate themselves.
Generalized Anxiety Disorder-7 (GAD-7) Turkish Form | Baseline, post-test (6 weeks later from baseline), follow up (10 weeks later from baseline)
  It will use for anxiety symptoms level. The GAD-7 consists of 7 items structured in a four-point Likert scale to measure anxiety level. The lowest score is 0 and the highest score is 21. A high score indicates a high level of anxiety. It is a self-report tool and participants evaluate themselves.

OTHER OUTCOMES:
Sociodemographic Information Form | Baseline
  This form will assess age, gender and whether the participant has received psychotherapy/counselling or medication before as potential covariates.
System Usability Scale (SUS-10) Turkish Form | Post-test (6 weeks later from baseline)
  This is a tool aiming to assess the impact of program usability on treatment outcomes. SUS-10 was developed to assess the usability of a system. It consists of 10 items. The items are on a 5-point Likert scale (0-4). The lowest score is 0 and the highest score is 40. A high score indicates high usability. Raw scores are multiplied by 2.5 when calculating. A score above 70 is considered as sufficient usability.
Attitudes Toward Internet-Based Interventions Scale (ETAM) Turkish Form | Baseline
  ETAM will use people's opinions/attitudes about internet-based interventions. It consists of 16 items. It is defined as a five-point Likert scale. A high score indicates a positive attitude towards internet-based interventions.
Adherence to Intervention | Post-test (6 weeks later from baseline)
  Adherence refers to the degree to which the user follows the program as designed. The calculation of adherence will use the percentage determined by dividing the number of core modules completed by the participant during the post-test by the total number of core modules in the program and multiplying it by 100.
Guide Evaluation | End of the experiment
  It is a one-question assessment in which the participants in the guided intervention group rate the feedback they received at the end of the program and their relationship with the guide. Participants will score their communication with the guide between 1-10 points.